CLINICAL TRIAL: NCT01673204
Title: Clinical Trial Technology Development for the Validation of Surrogate Prognostic Markers in Patients With Diabetic Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yon Su Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SNUH-TNFR
Record Dates: First submitted 2012-08-21; First posted 2012-08-27 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Diabetic Nephropathy
Keywords: surrogate marker,; circulating soluble TNF receptor,; diabetic nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Calcitriol (Experimental): Calcitriol
  Interventions: Drug: Calcitriol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitriol — dosage of 0.5mcg administered orally once daily for 12 month
  Arms: Calcitriol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Worldwide, the most common cause of chronic kidney disease (CKD) and end stage renal disease (ESRD) is diabetes. Unlike the past, in south korea, diabetes account for more than 40% of ESRD. According to WHO reports in 1998, 100 million people had type 2 diabetes in 1997, and there is expected to increase by 300 million people in 2025. In addition, the expected survival time of patients with diabetes increase compared to previous. In the future, ESRD due to type 2 diabetes is expected to have a significant impact on the health industry. Therefore, prevention of progression to CKD and ESRD in diabetic patients is important to aspect of national health and economic problems. How to stop the progression of diabetic nephropathy is part of modern medicine to be solved.

Strict glycemic control, blood pressure regulation, and use of renin-angiotensin system (RAS) blockers inhibit the development and progression of diabetic nephropathy. Microalbuminuria in diabetic patients has been recognized as a predictor of progression of diabetic nephropathy. Thus, the prevention of elevated urinary albumin excretion is an important therapeutic target for the prevention of renal and cardiovascular events.

In patients with diabetes and hypertension, the drugs that block the RAS are used to treat proteinuria, but still a large number of patients with proteinuria are uncontrolled. In addition, ACE inhibitors or ARB agents actually have a limited effect on reducing the risk of cardiovascular or renal outcome. Also, sulodexide or pentoxyphylline which is reducing proteinuria have some weak evidence in terms of efficacy and safety. Therefore, the introduction of new alternative drugs are required.

Already several study reported that calcitriol or paricalcitol in the renal injury model have renopreventive effect. In addition, in diabetic renal injury mice model reported that vitamin D receptor deficiency leads to glomerulosclerosis. Inhibition of the RAS with combination of paricalcitol and RAS inhibitors effectively prevent renal injury in diabetic nephropathy. Recently, Dick de Zeeuw et al reported that addition of paricalcitol to RAS inhibition safely lower residual albuminuria in patients with diabetic nephropathy. Recent studies reported that elevated concentrations of serum markers of the TNFα and Fas-pathways are strongly associated with decreased renal function in diabetic patients. However, the role of these markers in early progressive renal function decline are not clear. Therefore, the objective of this study is to identify the renoprotective effect as an new treatment of activated vitamin D (Calcitriol) indicating the TNF-α-related anti-inflammatory action and to seek the role as an important biomarker that the changes of TNFR in diabetic nephropathy can predict response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients age 19-80 years
* Clinically proven diabetic nephropathy
* MDRD eGFR >= 30mL/min/1.73m2
* Patients with residual urine protein/creatinine ratio >= 200mg/g
* Adequate blood pressure control as treated systolic blood pressure <=140 or diastolic <=90 mmHg with RAS inhibitor for more than 3months
* Serum intact PTH <500 mg/dL
* Serum calcium <10.2 mg/dL
* Patients who have not been treated vitamin D within the 3months prior to signing the informed consent form

Exclusion Criteria:

* Patients age <19 years or > 80years
* Patients with rapidly progressive glomerulonephritis
* Patients requiring renal replacement therapy immediately
* Hypercalcemia(Uncorrected serum calcium level >10.2 mg/dL) within recent 3month
* Malignant hypertension
* Heart failure (New York Heart Association functional class II to IV or LVEF <40%)
* Severe chronic obstructive lung disease
* Decompensated liver disease (ALT >3X upper normal limit)
* Known allergy or hypersensitivity to vitamin D
* Current treatment with steroids and/or immunosuppressive agents
* Active primary malignancy requiring treatment or survival limits less than 2years
* History of noncompliance to medical regimen
* Inability to give an informed consent or to cooperate with researchers

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Changes in renal function with proteinuria | 12 month after administration
  Comparison of in GFR level from baseline Comparison of proteinuria amount checked by random urine protein/creatinine ratio

SECONDARY OUTCOMES:
changes in sTNFR and TNF-related proteins | 12 months after administration
  Comparison of serum TNFR1, TNFR2 levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yonsu Kim, M.D., Ph.D, Study Chair — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul